CLINICAL TRIAL: NCT03638635
Title: TAP Blocks Performed With Bupivacaine Versus Liposomal Bupivacaine in Colorectal Surgery Patients: A Prospective, Cluster Randomized Trial
Brief Title: Standard Bupivacaine vs Liposomal Bupivacaine in Colorectal Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of personnel available to complete study.
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 17-2725
Record Dates: First submitted 2017-08-21; First posted 2018-08-20 (Actual); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-04

CONDITIONS: Opioid Use; Pain, Postoperative; Colectomy; Colorectal Surgery
Keywords: Bupivacaine; Exparel; TAP Block; Opioids; Narcotics; ERAS
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive either standard bupivacaine or liposomal bupivacaine.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and the floor nursing staff recording pain scores will be blinded to the assigned intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Bupivacaine (Active Comparator): Standard (0.25% bupivacaine) bupivacaine (133 mg in 10mL, diluted with 20 mL saline) will be injected into the fascial layer between the internal oblique and the transversus abdominis with ultrasound guidance, 30 mL per side for a total of 60 mL.
  Interventions: Drug: Bupivacaine
- Bupivacaine Liposome (Experimental): Liposomal bupivacaine (133 mg in 10mL, diluted with 20 mL saline) will be injected into the fascial layer between the internal oblique and the transversus abdominis with ultrasound guidance, 30 mL per side for a total of 60 mL.
  Interventions: Drug: Bupivacaine liposome

INTERVENTIONS:
Drug: Bupivacaine — Abdominal injection of bupivacaine into fascial layer.
  Other Names: Marcaine
  Arms: Standard Bupivacaine
Drug: Bupivacaine liposome — Abdominal injection of bupivacaine liposome into fascial layer.
  Other Names: Exparel
  Arms: Bupivacaine Liposome

SUMMARY:
The transversus abdominis plane (TAP) block can be used to reduce pain in patients who get abdominal surgery. TAP blocks are given with a local anesthetic. The purpose of this study is to compare pain medication usage after surgery between two different types of local anesthetic: liposomal bupivacaine and standard bupivacaine.

DETAILED DESCRIPTION:
Pain control is a factor that is central to the surgical patient's postoperative experience. Opioid pain medications are a mainstay of postoperative pain management. However, these have several adverse effects.

Multimodal pain regimens to minimize opioid use have become central to enhanced recovery after surgery (ERAS) protocols. The transversus abdominis plane (TAP) block is one intervention that contributes to this regimen. Traditionally, TAP blocks are performed with local anesthetics such as bupivacaine. More recently, these have also been performed with liposomal bupivacaine, whose duration of action is much greater than regular bupivacaine (96 hours versus 8-9 hours, respectively).

In this study, postoperative opioid usage will be compared between patients receiving regular bupivacaine and liposomal bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing elective colectomy by surgeons of Fairfax Colon and Rectal Surgery

Exclusion Criteria:

* Allergic to local anesthetics
* Unable to provide consent
* Pregnant
* On opioids at home chronically (Patients previously on a regular opioid regimen would need to be opioid-free for a period of 1 year for inclusion in the study)
* Undergoing emergent operations
* Undergoing loop ileostomy reversal
* Undergoing abdominoperineal resection, pelvic exenteration, or perineal rectal prolapse repairs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Colvin, MD, Principal Investigator — Inova Health Care System
Locations (6):
- United States (6):
  - Fairfax Colon & Rectal Surgery, Alexandria Office, Alexandria, Virginia
  - Fairfax Colon & Rectal Surgery, Fairfax-Prosperity Office, Fairfax, Virginia
  - Fairfax Colon & Rectal Surgery, Fair Oaks Office, Fairfax, Virginia
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Fairfax Colon & Rectal Surgery, Loudoun Office, Lansdowne Town Center, Virginia
  - Fairfax Colon & Rectal Surgery, Reston Office, Reston, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Background] Young MJ, Gorlin AW, Modest VE, Quraishi SA. Clinical implications of the transversus abdominis plane block in adults. Anesthesiol Res Pract. 2012;2012:731645. doi: 10.1155/2012/731645. Epub 2012 Jan 19. PMID 22312327
- [Background] Rashid A, Gorissen KJ, Ris F, Gosselink MP, Shorthouse JR, Smith AD, Pandit JJ, Lindsey I, Crabtree NA. No benefit of ultrasound-guided transversus abdominis plane blocks over wound infiltration with local anaesthetic in elective laparoscopic colonic surgery: results of a double-blind randomized controlled trial. Colorectal Dis. 2017 Jul;19(7):681-689. doi: 10.1111/codi.13578. PMID 27943522
- [Background] Oh TK, Yim J, Kim J, Eom W, Lee SA, Park SC, Oh JH, Park JW, Park B, Kim DH. Effects of preoperative ultrasound-guided transversus abdominis plane block on pain after laparoscopic surgery for colorectal cancer: a double-blind randomized controlled trial. Surg Endosc. 2017 Jan;31(1):127-134. doi: 10.1007/s00464-016-4941-7. Epub 2016 Apr 29. PMID 27129571
- [Background] Walter CJ, Maxwell-Armstrong C, Pinkney TD, Conaghan PJ, Bedforth N, Gornall CB, Acheson AG. A randomised controlled trial of the efficacy of ultrasound-guided transversus abdominis plane (TAP) block in laparoscopic colorectal surgery. Surg Endosc. 2013 Jul;27(7):2366-72. doi: 10.1007/s00464-013-2791-0. Epub 2013 Feb 7. PMID 23389068
- [Background] Favuzza J, Delaney CP. Outcomes of discharge after elective laparoscopic colorectal surgery with transversus abdominis plane blocks and enhanced recovery pathway. J Am Coll Surg. 2013 Sep;217(3):503-6. doi: 10.1016/j.jamcollsurg.2013.03.030. Epub 2013 Jun 28. PMID 23810575
- [Background] Ris F, Findlay JM, Hompes R, Rashid A, Warwick J, Cunningham C, Jones O, Crabtree N, Lindsey I. Addition of transversus abdominis plane block to patient controlled analgesia for laparoscopic high anterior resection improves analgesia, reduces opioid requirement and expedites recovery of bowel function. Ann R Coll Surg Engl. 2014 Nov;96(8):579-85. doi: 10.1308/003588414X13946184900921. PMID 25350178
- [Background] Barron KI, Lamvu GM, Schmidt RC, Fisk M, Blanton E, Patanwala I. Wound Infiltration With Extended-Release Versus Short-Acting Bupivacaine Before Laparoscopic Hysterectomy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2017 Feb;24(2):286-292. doi: 10.1016/j.jmig.2016.11.002. Epub 2016 Nov 14. PMID 27856385
- [Background] Morales R Jr, Mentz H 3rd, Newall G, Patronella C, Masters O 3rd. Use of abdominal field block injections with liposomal bupivicaine to control postoperative pain after abdominoplasty. Aesthet Surg J. 2013 Nov 1;33(8):1148-53. doi: 10.1177/1090820X13510720. Epub 2013 Nov 8. PMID 24214950
- [Background] Haas E, Onel E, Miller H, Ragupathi M, White PF. A double-blind, randomized, active-controlled study for post-hemorrhoidectomy pain management with liposome bupivacaine, a novel local analgesic formulation. Am Surg. 2012 May;78(5):574-81. doi: 10.1177/000313481207800540. PMID 22546131
- [Background] Knudson RA, Dunlavy PW, Franko J, Raman SR, Kraemer SR. Effectiveness of Liposomal Bupivacaine in Colorectal Surgery: A Pragmatic Nonsponsored Prospective Randomized Double Blinded Trial in a Community Hospital. Dis Colon Rectum. 2016 Sep;59(9):862-9. doi: 10.1097/DCR.0000000000000648. PMID 27505115
- [Background] Hutchins JL, Kesha R, Blanco F, Dunn T, Hochhalter R. Ultrasound-guided subcostal transversus abdominis plane blocks with liposomal bupivacaine vs. non-liposomal bupivacaine for postoperative pain control after laparoscopic hand-assisted donor nephrectomy: a prospective randomised observer-blinded study. Anaesthesia. 2016 Aug;71(8):930-7. doi: 10.1111/anae.13502. Epub 2016 May 30. PMID 27238859
- [Background] Stokes AL, Adhikary SD, Quintili A, Puleo FJ, Choi CS, Hollenbeak CS, Messaris E. Liposomal Bupivacaine Use in Transversus Abdominis Plane Blocks Reduces Pain and Postoperative Intravenous Opioid Requirement After Colorectal Surgery. Dis Colon Rectum. 2017 Feb;60(2):170-177. doi: 10.1097/DCR.0000000000000747. PMID 28059913

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were approached for consent in the hospital postoperatively to request the use of their data for research purposes.
Period: Initial Hospitalization
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Started | 39 | 24
Completed | 39 | 22
Not Completed | 0 | 2
Not completed — Study terminated prematurely | 0 | 1
Not completed — Withdrawal by study personnel | 0 | 1
Period: Follow-Up (30 Days After Discharge)
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Started | 39 | 22
Completed | 0 | 0
Not Completed | 39 | 22
Not completed — Study terminated prematurely | 39 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome | Total
Number analyzed (Participants) | 39 | 24 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.97 (16.25) | 60.04 (17.36) | 60.63 (16.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 13 | 35
  Male | 17 | 11 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 30 | 20 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 24 | 63

OUTCOME MEASURES:

1. Primary Outcome: In-hospital Postoperative Opioid Consumption
Description: Daily overall opioid use recorded as morphine equivalents
Time Frame: up to postoperative day 3 at 1 pm
Population: The amount of in-hospital postoperative opioid consumption was going to be obtained from the charts, where it is recorded as standard of care. However, this study was terminated prematurely before data could be collected from the charts; therefore no data are available for this outcome measure.
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Pain Score
Description: Recorded on a scale of 0 (No pain) to 10 (Worst possible pain)
Time Frame: Approximately every 6 hours through postoperative day 3 by 1 pm
Population: Outcome data reported for patients with non-missing data. Pain scores presented are the first postoperative pain score per subject only due to missing data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Number analyzed (Participants) | 37 | 21
units on a scale | 3 [0 to 5] | 3 [0 to 6]

3. Secondary Outcome: Time to Patient Mobilization
Description: Number of days from day of surgery until patient mobilization
Time Frame: From time of surgery until time of first patient ambulation post op. Assessed until date of discharge (usually up to 4 days after surgery).
Population: Outcome data reported for subjects with non-missing data.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Number analyzed (Participants) | 29 | 18
days | 1 [0 to 1] | 0.5 [0 to 1]

4. Secondary Outcome: Time to Return of Bowel Function
Description: Number of days from time of surgery until return of bowel function
Time Frame: From time of surgery until first time patient passes gas or stool per rectum or into ostomy bag. Assessed until date of discharge (usually up to 4 days after surgery).
Population: Outcome data reported for subjects with non-missing data.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Number analyzed (Participants) | 28 | 18
days | 2 [1 to 2] | 2 [1 to 2]

5. Secondary Outcome: Time to Clear Liquid Diet
Description: Number of days from time of surgery until patient tolerates clear liquid diet
Time Frame: From time of surgery until first time patient tolerates clear liquids without nausea or vomiting. Assessed until date of discharge (usually up to 4 days after surgery).
Population: Outcome data reported for subjects with non-missing data.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Number analyzed (Participants) | 29 | 18
days | 0 [0 to 0] | 0 [0 to 1]

6. Secondary Outcome: Time to Low Fiber Diet
Description: Number of days from day of surgery until patient tolerates low fiber diet
Time Frame: From time of surgery until first time patient tolerates a low fiber diet without nausea or vomiting. Assessed until date of discharge (usually up to 4 days after surgery).
Population: Outcome data reported for subjects with non-missing data.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Number analyzed (Participants) | 28 | 17
days | 1.5 [1 to 2.25] | 1 [1 to 3]

7. Secondary Outcome: Length of Stay
Description: Total postoperative hospital stay in days
Time Frame: Date of surgery to date of discharge (usually up to 4 days after surgery).
Population: Outcome data reported for subjects with non-missing data.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Number analyzed (Participants) | 31 | 18
days | 3 [3 to 5] | 3.5 [3 to 5.75]

8. Secondary Outcome: In-hospital Antiemetic Use
Description: Amount of ondansetron patient required postoperatively during hospital stay, in milligrams
Time Frame: Time of transfer to post operative suite to time of discharge (usually up to 4 days after surgery).
Population: Outcome data reported for subjects with non-missing data.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Number analyzed (Participants) | 31 | 17
mg | 2.9 (3.6) | 5.6 (12.5)

9. Secondary Outcome: Complications
Description: Patient suffered a complication (infection, small bowel obstruction, dehydration, deep vein thrombosis/pulmonary embolism, anastomotic leak, cardiac arrest, stroke, sepsis) after surgery
Time Frame: Within 30 days of surgery
Population: Complications data was going to be collected from chart review. However, the study was prematurely terminated before this data could be collected.
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Readmissions
Description: Patient readmitted to hospital after discharge
Time Frame: Within 30 days of hospital discharge
Population: Readmissions data was going to be collected from chart review. However, the study was prematurely terminated before this data could be collected.
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Mortality
Description: Patient death after surgery
Time Frame: Within 30 days of surgery
Population: Mortality data was going to be collected from chart review. However, the study was prematurely terminated before this data could be collected.
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Hospitalization Costs
Description: Total hospitalization costs per patient per this surgical encounter
Time Frame: From date of this surgical admission to date of this surgical discharge (usually up to 4 days after surgery).
Population: Cost data was intended to be collected through the finance department at the end of the study. However, the study was terminated prematurely, so cost data is not able to be obtained.
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days post-enrollment
Arm/Group | Standard Bupivacaine | Bupivacaine Liposome
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/24
Other Adverse Events (participants affected / at risk) | 0/39 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Bupivacaine (N=39) | Bupivacaine Liposome (N=24)
Hospitalization (Surgical and medical procedures) | 0 (0) | 1 (1) — Return to the operating room

LIMITATIONS AND CAVEATS:
Early termination due to lack of resources leading to incomplete data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT03638635/Prot_SAP_000.pdf